CLINICAL TRIAL: NCT00309244
Title: A Prospective, Multi-Center, Open-Label, Randomized, Controlled Clinical Trial Comparing the Efficacy and Safety in Subjects With Type 2 Diabetes Receiving Subcutaneous Basal Insulin and Prandial Inhalation of Technosphere /Insulin Versus Subcutaneous Premixed Insulin Therapy Over a 52-Week Treatment Period and a 4-Week Follow-up
Brief Title: Efficacy and Safety in Subjects With Type 2 Diabetes Receiving Subcutaneous Basal Insulin and Prandial Inhalation of Technosphere/Insulin Versus Subcutaneous Premixed Insulin Therapy Over a 52-Week Treatment Period and a 4-Week Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MKC-TI-102
Record Dates: First submitted 2006-03-27; First posted 2006-03-31 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

ARMS (2):
- TI + Insulin glargine (Experimental): Technosphere® Insulin Inhalation Powder + insulin glargine
  Interventions: Drug: Technosphere® Insulin Inhalation Powder
- BPR 70/30 (Active Comparator): 70% insulin aspart protamine suspension and 30% insulin aspart injection (rDNA origin)
  Interventions: Drug: 70% insulin aspart protamine suspension and 30% insulin aspart injection (rDNA origin)

INTERVENTIONS:
Drug: Technosphere® Insulin Inhalation Powder — Inhalation, 15U/30U
  Arms: TI + Insulin glargine
Drug: 70% insulin aspart protamine suspension and 30% insulin aspart injection (rDNA origin) — BPR 70/30, which is a premix of intermediate acting and rapid acting insulin given sc
  Arms: BPR 70/30

SUMMARY:
The purpose of this 13 month study (12 month treatment period and 1 month follow-up period) is to determine whether inhaled insulin is safe and effective in the treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 80 years old
* Clinical diagnosis of type 2 diabetes mellitus
* HbA1c > 7.0% and ≤ 11.0%
* BMI ≤ 40 kg/m2
* Negative smoking status and urine cotinine test
* Written informed consent
* Receiving sc insulin 2-3 times daily administered as any of the following 3 regimens: self-mix regimen, pre-mix regimen, or long-acting analogue and regular or rapid-acting insulin analogue not to exceed 3 daily injections. Subjects may also have received oral antidiabetic agents including metformin or thiazolidinediones.
* No dose adjustments for insulin and oral antidiabetic agents within the preceding 6 weeks.
* FEV1 ≥ 70% of NHANES III predicted; TLC) ≥ 80% of predicted (Intermountain Thoracic Society); DLCO uncorrected ≥ 70% of predicted

Exclusion Criteria:

* Total daily dose of insulin ≥1.4 IU/kg body weight
* Treatment with any sulfonylureas and/or meglitinides and/or alpha-glucosidase inhibitors within the preceding 8 weeks
* Treatment with pramlintide acetate (Symlin®), and/or any incretins (e.g., exenatide [Byetta®]) within the preceding 8 weeks
* Unstable diabetes mellitus control, defined as 2 or more episodes of severe hypoglycemia (requiring third party intervention) and/or any hospitalization or emergency room visit due to poor diabetic control or hyperglycemia requiring hospitalization within the preceding 6 months
* Exposure to an inhaled insulin at any time, treatment with an investigational drug within the preceding 3 months, and/or current participation in another clinical trial
* Allergy to insulin or to any drugs to be used as part of the clinical trial, or history of hypersensitivity to the investigational drug or to drugs of similar chemical structures
* History of active viral and/or cirrhotic hepatic disease and/or abnormal liver enzymes as evidenced by serum aspartate aminotransferase (AST)and/or alanine aminotransferase (ALT) ≥ 3 x Upper Limit of Normal (ULN)(Includes active hepatitis A, positive hepatitis B and/or hepatitis C serology)
* Serum creatinine > 1.8 mg/dL in women and > 2.0 mg/dL in men History of chronic obstructive pulmonary disease (COPD), asthma (any history of bronchospasm or asthma after the age of 14), and/or any other clinically important pulmonary disease confirmed by documented history, pulmonary function testing, or radiologic findings
* Congestive heart disease graded as class III or class IV according to New York Heart Association criteria and subjects currently being treated pharmacologically for ventricular dysrhythmias using amiodarone
* History of myocardial infarction, cardiac surgery, coronary angioplasty, and/or stroke within the preceding 3 months
* Symptomatic coronary artery disease, including crescendo angina, unstable angina, and/or unstable or symptomatic cardiac arrhythmias
* Poorly controlled arterial hypertension despite pharmacologic treatment, defined as systolic blood pressure (BP) > 180 mm Hg and/or diastolic BP > 110 mm Hg at screening
* History of malignancy within the preceding 5 years (other than excised basal cell carcinoma of the skin), any history of lung neoplasm, and/or subjects with current or previous chemotherapy or radiation therapy that may result in pulmonary toxicity
* History of acquired immunodeficiency syndrome (AIDS), AIDS-related complex (ARC), or positive human immunodeficiency virus (HIV) serology
* Prior diagnosis of systemic autoimmune or collagen vascular disease requiring previous or current treatment with systemic corticosteroids, cytotoxic drugs, or penicillamine
* Visit 1/Screening (Week -3), but prior to Visit 1 PFTs and before Visit 3/Baseline (Week 0), subject will be scheduled for PFTs after 30 days from resolution of respiratory infection. An additional hemoglobin and urine β-HCG (for women of childbearing potential age only) will be required
* Women who are pregnant, lactating or planning to become pregnant
* Women of childbearing potential (defined as pre-menopausal and not surgically sterilized or postmenopausal for less than 2 years) not practicing adequate birth control. Adequate birth control is defined as using oral, percutaneous and/or transdermal contraceptives; condoms and diaphragms with a spermicide, or intrauterine devices
* Current drug and/or alcohol abuse
* Subjects who in the opinion of the Investigator will be unable to comply with the requirements of the protocol
* Severe complications of diabetes mellitus, in the opinion of the Investigator, including: symptomatic autonomic neuropathy, disabling peripheral neuropathy, active proliferative retinopathy; nephropathy with renal failure, renal transplant and/or dialysis; history of foot ulcers; nontraumatic amputations due to gangrene;and/or vascular claudication
* Any other concurrent medical or major psychiatric condition which, in the opinion of the Investigator, makes the subject unsuitable for the clinical trial, or could limit the validity of the ICF and/or impair the subject's ability to participate in the trial
* Inability to perform PFT maneuvers meeting recommended American Thoracic Society (ATS) acceptability and repeatability criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2006-02; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (151):
- United States (80):
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Quality of Life Medical & Research Center, Tucson, Arizona
  - Southern Arizona VA Healthcare System, Tucson, Arizona
  - Tucson Clinical Research, Tucson, Arizona
  - International Clinical Research Network, Chula Vista, California
  - Saad Hijazi MD Inc, Fresno, California
  - Valley Research, Fresno, California
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - South Bay Clinical Research, Inglewood, California
  - Southern California Endocrine Center, Pasadena, California
  - Coastal Biomedical Research Inc, Santa Monica, California
  - Diabetes Research Center, Tustin, California
  - University of Miami Diabetes Research Institute, Miami, Florida
  - International Research Associates LLC, Miami, Florida
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Atlanta Pharmaceutical Research Center, Dunwoody, Georgia
  - North Atlanta Endocrinology & Diabetes PC, Lawrenceville, Georgia
  - Atlanta Center for Clinical Research, Roswell, Georgia
  - John H Stoger Jr Hospital of Cook County, Chicago, Illinois
  - Clintell Inc, Skokie, Illinois
  - Clintell Inc (Ellyin), Skokie, Illinois
  - Medical Research of Louisiana, Metairie, Louisiana
  - Joslin Diabetes Center University of Maryland Medicine, Baltimore, Maryland
  - James A Dicke MDPA, Towson, Maryland
  - Wayne State University, Detroit, Michigan
  - Michigan Institute of Medicine, Livonia, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - Radiant Research Inc (Minneapolis), Edina, Minnesota
  - International Diabetes Center, Minneapolis, Minnesota
  - Center for Urologic Clinical Trials University of Minnesota, Minneapolis, Minnesota
  - Amin Radparvar's Private Practice, City of Saint Peters, Missouri
  - MedEx Healthcare Research Inc, St Louis, Missouri
  - Billings Clinic Research Division, Billings, Montana
  - Montana Health Research Institute, Billings, Montana
  - Creighton Diabetes Center, Omaha, Nebraska
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - University of New Mexico HCS, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Univeristy of Physicians Group Endocrine Division, Staten Island, New York
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - East Carolina University (Tanenberg), Greenville, North Carolina
  - Physician's East PA, Greenville, North Carolina
  - Valley Medical Primary Care, Centerville, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Health Partners - Center of Clinical Research, Dayton, Ohio
  - Cleveland Clinic Health System, East Cleveland, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Oregon Medical Group Clinical Resesarch, Eugene, Oregon
  - Lane Medical Research Group, Eugene, Oregon
  - Portland Diabetes & Endocrinology Center, Portland, Oregon
  - New Hope Research of Oregon, Portland, Oregon
  - Covance CRU Inc., Portland, Oregon
  - Pennsylvania Research Institute, Bensalem, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Southeastern Research Associates Inc, Taylors, South Carolina
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Memphis Internal Medicine PLLC, Memphis, Tennessee
  - The Endocrine Clinic, Memphis, Tennessee
  - Israel Hartman MD, Arlington, Texas
  - South Arlington Primary Care Assoc PA, Arlington, Texas
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Radiant Research Dallas-North, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - Spuhler Medical Associates, Friendswood, Texas
  - Clinical Trial Network, Houston, Texas
  - Quality Assurance Research Center Inc, San Antonio, Texas
  - Covenant Clinic Research, San Antonio, Texas
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Sentara Medical Group, Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Larry D Stonesifer MD Inc PS, Federal Way, Washington
  - Rainier Clinical Research Center Inc, Renton, Washington
  - Cedar Research, Tacoma, Washington
  - Liberty Research Center, Tacoma, Washington
- Argentina (7):
  - Hospital Interzonal de Agudos Pedro Fiorito, Avellaneda, Buenos Aires
  - CITDEEM - Centro de Investigacion y Tratamiento En Diabetes y Enfermedades Endocrino-Metabolicas, San Miguel de Tucumán, Tucumán Province
  - FUNDAPRES/CIMel, Buenos Aires
  - Centro Endocrinologic Tiempo, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Cons Asoc de Endocrinologia, Buenos Aires
  - Centro Medico Dra De Salvo, Buenos Aires
- Brazil (12):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - CPClin-Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - Universidade Estabual de Maringa, Maringa Parana
  - Nucleo de Medicina Integrada, Mogi das Cruzes
  - Instituto Estadual De Diabetes e Endocrinologia Luis Capriglione, Rio de Janeiro
  - Ccbr Brasil Centro de Analises e Pesquisas Clinicas Ltda, Rio de Janeiro
  - Hospital Guilherme Alvaro, Santos
  - Hospital do Rim e Hipertensao, São Paulo
  - Instituto da Saude e Bem Estar da Mulher, São Paulo
  - Blumenau Servicos Medicos S/C Ltda, São Paulo
  - Centro de Pesquisa Clinica e Medicina Avancada, São Paulo
- Canada (6):
  - Keele Medical Place, Downsview, Ontario
  - Quest Clinical Trials, Markham, Ontario
  - Lifestyle Metabolism Center, Oakville, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Lifestyle Metabolism Center, Thornhill, Ontario
  - Lifestyle Metabolism Center, Toronto, Ontario
- Chile (4):
  - Hospital del Salvador, Santiago, Santiago Metropolitan
  - Hospital Padre Alberto Hurtado, Santiago, Santiago Metropolitan
  - Hospital Clinico Pontificia Universidad Catolica de Chile, Santiago
  - Hospital San Borja ArriaranUniversidad de Chile, Santiago
- Mexico (6):
  - Instituto Mexicano de Investigacion, Mexico City, Durango
  - Hospital OCA, Monterrey, Nuevo Leon, MX
  - Hospital Universitario Dr Jose E Gonzalez, Monterrey, Nuevo León
  - Hospital Santa Engracia-CIMA, Garza García
  - Centro de Estudios en Diabetes, Mexico City
  - Cifbiotec, Mexico City
- Poland (7):
  - Oddzial Chorob Wewnetrznych, Bialystock, POL
  - NZOZ Specjalistyczny Osrodek Internistyczno - Diabetologiczny, Bialystok, POL
  - Katedra I Klinika Chorob Metabolicznych Collegium Medicum Uniwersytety Jagiellonskiego, Krakow, POL
  - Klliniczny nr 1 im Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz, POL
  - Instytut Centrum Zdrowia (009) Matki Polki, Lodz, POL
  - Szpital Kolejowy im Dr w Roeflera(009) Oddzial Gastorenterologii, Pruszków, POL
  - NZOZ Diabetologiczna Poradnia Specjalistyczna, Warsaw
- Russia (16):
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - NI Principal Military Clinical Hospital n a academician N.N. Burdenko of the Ministry of Defense, Moscow, RUS
  - NEI HPE Moscow State University of Medicine and Dentistry of FAHSD City Clinical Hospital #70, Moscow, RUS
  - Moscow City Clinical Hospital # 13, Moscow, RUS
  - SEI HPE Moscow Medical Academy IM Sechenov of Roszdrav Clinic of Endocrinology, Moscow, RUS
  - SI Internal Affairs of Moscow- Clinical Hospital, Moscow, RUS
  - RAAMS Endocrinology and Diabetology Department, Moscow, RUS
  - St Petersburg NHI City Polytclinic #77 City Diabetological Center #4, Saint Petersburg, RUS
  - Central Medical Sanitary Unit #122, Saint Petersburg, RUS
  - Pavlov State Medical Univ of St Petersburg, Saint Petersburg, RUS
  - NEI HPE Smolensk State Medical Academy of FAHSD RNHI Smolensk Regional Clinical Hospital, Smolensk, RUS
  - MHI Clinical Hospital for Emergency Care na NV Soloviev, Yaroslavl, RUS
  - MCHI Medical Sanitary Unit of Novo-Yaroslavsky Oil Refining Plant, Yaroslavl, RUS
  - NHI Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - NI Central Clinical Hospital of RAS, Moscow
  - City Clinical Hospital # 61, Moscow
- Spain (9):
  - Complejo Hospitalario Nuestra Senora de Valme, Seville, Andalusia
  - Hospital de Mataro, Mataró, Barcelona
  - Hospital del Mar (Cano), Barcelona
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario de la Princessa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Corporacion Sanitaria Parc Tauli Unidad de Endocrinologia, Sabadell
  - Complejo Hospitalario Virgen del Rocio, Seville
  - Hospital Virgen Macarena (policlinico) 2ª planta Servicio de Endocrinologia y Nutricion, Seville
- United Kingdom (4):
  - Birchwood Surgery, Letchworth Garden City, Herts
  - Lister Hospital, Stevenage, Herts
  - Guy's & St Thomas Hospital, London
  - Yaxley Group Practice, Peterborough

REFERENCES:
- [Derived] Peyrot M, Rubin RR. Patient-reported outcomes in adults with type 2 diabetes using mealtime inhaled technosphere insulin and basal insulin versus premixed insulin. Diabetes Technol Ther. 2011 Dec;13(12):1201-6. doi: 10.1089/dia.2011.0037. Epub 2011 Oct 14. PMID 21999640
- [Derived] Rosenstock J, Lorber DL, Gnudi L, Howard CP, Bilheimer DW, Chang PC, Petrucci RE, Boss AH, Richardson PC. Prandial inhaled insulin plus basal insulin glargine versus twice daily biaspart insulin for type 2 diabetes: a multicentre randomised trial. Lancet. 2010 Jun 26;375(9733):2244-53. doi: 10.1016/S0140-6736(10)60632-0. PMID 20609970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled Feb. 23, 2006 Multi-national trial conducted in US, Canada, Mexico, Brazil, Argentina, Chile, Spain, UK, Poland, Russia
Pre-assignment Details: 3 week Screening period prior to randomization - 2064 Screened / 673 Eligible . 677 subjects were randomized. ( 4 ineligible subjects were randomized in error) 1391 screen failures.
  23 Subjects randomized but never dosed.
Groups:
- TI + Insulin Glargine: Technosphere® Insulin Inhalation Powder (administered at each meal) + subcutaneous insulin glargine (administered once daily at bedtime). Doses are individualized for each patient.
- BPR 70/30: 70% insulin aspart protamine suspension and 30% insulin aspart subcutaneous injection (rDNA origin), administered twice daily (before breakfast and before main evening meal). Doses are individualized for each patient.
Period: Overall Study
Arm/Group | TI + Insulin Glargine | BPR 70/30
Started | 334 | 343
Completed | 216 | 246
Not Completed | 118 | 97
Not completed — Adverse Event | 29 | 12
Not completed — Lost to Follow-up | 6 | 22
Not completed — Physician Decision | 5 | 8
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal by Subject | 50 | 32
Not completed — Various | 7 | 7
Not completed — Randomized but not dosed | 11 | 12
Not completed — Death | 4 | 1

BASELINE CHARACTERISTICS:
Population: Safety population (23 Subjects randomized but never dosed are not included).
Groups:
- Total: Total of all reporting groups
Arm/Group | TI + Insulin Glargine | BPR 70/30 | Total
Number analyzed (Participants) | 323 | 331 | 654
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.68) [19 to 79] | 55.9 (9.91) [24 to 78] | 55.9 (10.29) [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 185 | 345
  Male | 163 | 146 | 309
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: milligrams per deciliter] — TI + Insulin glargine arm,302 subjects BPR 70/30 arm, 316 subjects
  milligrams per deciliter | 171.8 (68.53) | 176.2 (67.15) | 174 (67.82)
HbA1c [Mean (Standard Deviation); unit: percentage] — Glycosylated Hemoglobin
  percentage | 8.7 (1.14) | 8.7 (1.10) | 8.7 (1.12)
Weight [Mean (Standard Deviation); unit: kilogram] — Weight in kg TI + Insulin glargine arm, 322 subjects BPR 70/30 arm, 331 subjects
  kilogram | 88.1 (17.33) | 85.7 (18.07) | 86.9 (17.74)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c to Week 52
Time Frame: Baseline to Week 52
Population: Intention to treat (ITT) with Last Observation Carried Forward (LOCF); participants with available data at baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 302 | 316
percent | -0.59 (0.063) | -0.71 (0.061)
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; Test type: Non-Inferiority or Equivalence — Sample size was set to meet regulatory requirement of 250 subjects per arm with 52-week data, resulting in > 90% power for a non-inferiority test of the difference in 12-month change of HbA1c scores between treatment groups with non-inferiority margin of 0.4%, standard deviation of 1.2 and 1-sided alpha of 0.025. Allowing for a 25% drop-out rate, 677 subjects were randomized; ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.05 to 0.29], Standard Error of Mean 0.085

2. Secondary Outcome: Change From Baseline in Weight to Week 52
Time Frame: Baseline to Week 52
Population: Intention to treat (ITT) population; participants with available data at baseline and Week 52.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 194 | 227
kilogram | 0.9 (0.32) | 2.5 (0.29)
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; ANCOVA model with terms of pooled site and treatment as fixed effects and baseline weight as covariate; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Net) = -1.6, 95% CI 2-sided [-2.4 to -0.7], Standard Error of Mean 0.41

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose to Week 52
Time Frame: Baseline to Week 52
Population: Intention to treat (ITT) population; participants with available data at baseline and Week 52.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 197 | 218
milligrams per deciliter | -35.7 (4.61) | -17.9 (4.21)
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; ANCOVA model with terms of pooled site and treatment as fixed effects and baseline fasting plasma glucose as covariate; Test type: Superiority or Other; p = 0.0029, ANCOVA; Mean Difference (Net) = -17.7, 95% CI 2-sided [-29.3 to -6.1], Standard Error of Mean 5.90

4. Secondary Outcome: Number of Subjects Achieving Week 52 HbA1c Levels Less Than or Equal to 7.0%
Time Frame: Week 52
Population: Intention to treat (ITT); participants with available data at baseline and Week 52.
Measure: Number; unit: participants
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 213 | 243
participants | 47 | 65
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; logistic regression analysis with the terms of treatment and baseline HbA1c in the model; Test type: Superiority or Other; p = 0.2793, Regression, Logistic; Odds Ratio (OR) = 0.774, 95% CI 2-sided [0.486 to 1.231]

5. Secondary Outcome: Incidence of Total Hypoglycemia
Description: Defined as hypoglycemic symptoms that are relieved with carbohydrate intake or blood glucose measurement <= 63 mg/dL, regardless of symptoms.
Time Frame: 52 Weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 323 | 331
percentage of participants | 47.99 | 68.58
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.423, 95% CI 2-sided [0.307 to 0.581] — Model: Treatment + Site

6. Secondary Outcome: Incidence of Severe Hypoglycemia
Description: Severe hypoglycemia occurs when all 3 of the following occur simultaneously:
  * Subject requires the assistance of another person;
  * Subject exhibits at least 1 cognitive neurological symptom (memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, seizure, loss of consciousness);
  * Measured BG is ≤ 49 mg/dL (2.7 mmol/L), or, in the absence of a BG measurement, clinical symptoms are reversed by oral carbohydrates, sc glucagon or intravenous glucose administration; OR,
  * Measured BG is ≤ 36 mg/dL (2.0 mmol/L) with or without symptoms.
Time Frame: 52 Weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 323 | 331
percentage of participants | 4.33 | 9.97
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; Test type: Superiority or Other; p = 0.0066, Regression, Logistic; Odds Ratio (OR) = 0.409, 95% CI 2-sided [0.215 to 0.780] — Model: Treatment + Site

7. Secondary Outcome: Total Hypoglycemia Event Rate
Description: Number of Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: 52 Weeks
Population: Safety Population
Measure: Number; unit: Number of events/subject-month
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 323 | 331
Number of events/subject-month | 0.41 | 0.61
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; Test type: Superiority or Other; p = 0.0027, Generalized Estimation Equation; Based on Poisson distribution

8. Secondary Outcome: Severe Hypoglycemia Event Rate
Description: Number of Severe Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: 52 Weeks
Population: Safety Population
Measure: Number; unit: Number of events/100 subject-months
Arm/Group | TI + Insulin Glargine | BPR 70/30
Number analyzed (Participants) | 323 | 331
Number of events/100 subject-months | 0.73 | 2.20
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs BPR 70/30; Test type: Superiority or Other; p = 0.0591, Generalized Estimating Equation; Based on Poission distribution

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after last dose
Arm/Group | TI + Insulin Glargine | BPR 70/30
Serious Adverse Events (participants affected / at risk) | 37/323 | 31/331
Other Adverse Events (participants affected / at risk) | 225/323 | 251/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TI + Insulin Glargine (N=323) | BPR 70/30 (N=331)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery atherosclerosis (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Optic atrophy (Eye disorders) | 0 | 1
Optic neuropathy (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Autoimmune disorder (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2
Diabetic foot infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 6
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TI + Insulin Glargine (N=323) | BPR 70/30 (N=331)
Upper respiratory tract infection (Infections and infestations) | 39 | 24
Nasopharyngitis (Infections and infestations) | 30 | 28
Influenza (Infections and infestations) | 18 | 18
Urinary tract infection (Infections and infestations) | 10 | 21
Hypoglycaemia (Metabolism and nutrition disorders) | 155 | 228
Headache (Nervous system disorders) | 18 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 106 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multi-center Study publication, PI may publish the Study results subject to MNKD rights herein.